CLINICAL TRIAL: NCT05187988
Title: Comparative Study Between Two Different Approaches of Brachial Plexus Block: Supraclavicular Approach and Retroclavicular Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Adel Mahmoud, resident doctor at anasthesia department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-11-02
Record Dates: First submitted 2021-11-28; First posted 2022-01-12 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Brachial Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular approach group (Active Comparator): probe placed firmly over the supraclavicular fossa, parallel to the clavicle to obtain a short-axis view of the divisions of the brachial plexus and the subclavian artery, lying on the first rib After skin infiltration with lidocaine 2% a 23-gauge 70mm block needle inserted in-plane with the ultrasound beam, in a lateral-to-medial direction, until the needle tip's positioned at the junction of the first rib and subclavian artery
  Interventions: Procedure: supraclavicular brachial plexus block
- Retroclavicular approach group (Active Comparator): the probe will be placed below and perpendicular to the clavicle, in a paramedian sagittal plane, medial to the coracoid process, to obtain a short-axis view of the cords of the brachial plexus and the axillary vessels. The needle will be then inserted in the supraclavicular fossa, approximately 1 cm posteriorly to the clavicle, and advanced in plane and strictly parallel to the ultrasound transducer. After passing the initial blind zone of about 2 cm caused by the acoustic shadow of the clavicle, the needle tip is constantly seen, until it is positioned posterior to the axillary artery
  Interventions: Procedure: Retroclavicular brachial plexus block

INTERVENTIONS:
Procedure: supraclavicular brachial plexus block — group will receive brachial plexus block above clavicle,Injection of anaesthetic will be done in brachial plexus around subclavian artery
  Arms: Supraclavicular approach group
Procedure: Retroclavicular brachial plexus block — group will receive brachial plexus block inferior to the clavicle,injection of anaesthetic will be done around axillary artery
  Arms: Retroclavicular approach group

SUMMARY:
In this study investigators will compare two different approaches of brachial plexus block ;supraclavicular approach and retroclavicular approach regarding success rate, duration of block, complications

ELIGIBILITY:
Inclusion Criteria:

* 100 patients doing distal arm surgery, elective , 18 to 60 years old , will be included in double blinded randomized study.

Exclusion Criteria:

* Patient refusal .
* local infection or deformity at the block site.
* Patient with significant neurological , psychiatric or neuromuscular disease.
* Pregnancy or lactating women .
* Coagulopathy .
* Morbid obesity .
* History of allergy to local anaesthetics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Block success rate | one year
  Investigator will compare success rate of both types of block and which one is more likely to be successfully administrated
Complications | one year
  Investigators will compare complications like pneumothorax,nerve injury,bleeding and which one is more likely to cause complications
Duration of sensory and motor blockade | one year
  Time which each procedure will take to block sensory and motor stimuli

SECONDARY OUTCOMES:
Duration of procedure | one year
  Time which took the investigator to administrate each type of block
Number of needle passes | one year
  number of times in which needle has entered been entered into the participant in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Albrecht E, Mermoud J, Fournier N, Kern C, Kirkham KR. A systematic review of ultrasound-guided methods for brachial plexus blockade. Anaesthesia. 2016 Feb;71(2):213-27. doi: 10.1111/anae.13347. Epub 2015 Dec 16. PMID 26670119
- [Background] Yazer MS, Finlayson RJ, Tran DQ. A randomized comparison between infraclavicular block and targeted intracluster injection supraclavicular block. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):11-5. doi: 10.1097/AAP.0000000000000193. PMID 25478758
- [Background] Charbonneau J, Frechette Y, Sansoucy Y, Echave P. The Ultrasound-Guided Retroclavicular Block: A Prospective Feasibility Study. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):605-9. doi: 10.1097/AAP.0000000000000284. PMID 26222346
- [Background] Grape S, Pawa A, Weber E, Albrecht E. Retroclavicular vs supraclavicular brachial plexus block for distal upper limb surgery: a randomised, controlled, single-blinded trial. Br J Anaesth. 2019 Apr;122(4):518-524. doi: 10.1016/j.bja.2018.12.022. Epub 2019 Jan 31. PMID 30857608